CLINICAL TRIAL: NCT03205800
Title: The Use of Temporary Anchorage Devices for Ridge Preservation After Tooth Extraction
Brief Title: Temporary Anchorage Devices for Ridge Preservation
Acronym: TAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Se-Lim Oh, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00076020
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Ridge Preservation

STUDY DESIGN:
Intervention Model Description: a split-mouth design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mini-screw placement (Experimental): One mini-screw (8 mm length) will be placed at the buccal plate of the extraction socket one week after the atraumatic extraction of maxillary first or second premolars in one side.
  Interventions: Device: Mini-screw
- No treatment (No Intervention): No treatment will be conducted on the contralateral side.

INTERVENTIONS:
Device: Mini-screw — Placement of a mini-screw
  Arms: Mini-screw placement

SUMMARY:
Alveolar bone is a bony portion surrounding the root of a tooth. The alveolar bone disappears gradually when the tooth is extracted. This bone loss often becomes a problem if a patient wants to close the missing tooth space with orthodontic treatments (braces), or to get a dental implant (a metal post replacing a tooth). Therefore, we would like to place small screws at the extraction sites to preserve the alveolar bone when the teeth need to be extracted and a patient cannot start treatments some time.

Mini-screws (small metal screws) are routinely used for regular orthodontic treatment. We will recruit patients who require extractions of two upper small molars (maxillary premolars) on both right and left sides. We will place one mini-screw on one side while the other side will be untouched after teeth extractions. Both sides will be followed at 8 months for examinations.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of transcortical mini-screws on ridge preservation following tooth extraction with a split mouth design. The study will evaluate clinical and radiographic outcomes following transcortical screw placements at extraction sites compared to non-treated extraction sites.

Specific Aim 1: To evaluate the clinical outcomes between the treated sites with a transcortical screw (the experimental group) and the non-treated sites (the control group) Null Hypothesis: There will be no differences in clinical parameters between the two groups.

Approach: The investigators will conduct a prospective split-mouth design clinical study. The investigators will compare the clinical changes in vertical bone height and horizontal bone width at 8 months from baseline (tooth extraction).

Specific Aim 2: To evaluate the radiographic outcome between the experimental group and the control group Null Hypothesis: There will be no difference in alveolar ridge height and width between the two groups.

Approach: The study will measure ridge height and width using cone beam computed tomography (CBCT) at baseline and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* two maxillary premolars (left and right) required to be extracted based on recommended dental treatment plans

Exclusion Criteria:

* uncontrolled hypertension
* diabetes mellitus
* subjects with a history of a long-term use of corticosteroid (> 6 months)
* subjects with a history of taking oral/IV bisphosphonates within the past 2 years
* smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Se-Lim Oh, Study Chair — University of Maryland School of Dentistry
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. The results will be published.

REFERENCES:
- [Derived] Joseph S, Oh SL, Pae EK, Joshi S. Use of transcortical miniscrews for alveolar ridge preservation following tooth extraction: A pilot study. Clin Oral Implants Res. 2022 Feb;33(2):150-157. doi: 10.1111/clr.13875. Epub 2021 Nov 16. PMID 34741321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study protocol was approved in October 2017 by the IRB. The recruitment period was from 1/12/2018 to 12/10/2018 at the University of Maryland Dental Clinics.
Pre-assignment Details: There was no significant event in this study that occur after participant enrollment and prior to assignment. One participant has both experimental (mini-screw placement) and control (no treatment) sides.
Units Other Than Participants: extraction site
Groups:
- No Treatment: No treatment will be conducted for extraction sockets on the contralateral side.
Period: Overall Study
Arm/Group | Mini-screw Placement | No Treatment
Started | 3; 6 extraction site | 3; 6 extraction site
Completed | 3; 6 extraction site | 3; 6 extraction site
Not Completed | 0; 0 extraction site | 0; 0 extraction site

BASELINE CHARACTERISTICS:
Population: Each participant contributed 2 units.
Units Other Than Participants: Teeth
Groups:
- No Treatment: No treatment will be conducted for the extraction site on the contralateral side.
- Total: Total of all reporting groups
Arm/Group | Mini-screw Placement | No Treatment | Total
Number analyzed (Participants) | 3 | 3 | 6
Number analyzed (Teeth) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (21) | 37 (21) | 37 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
Width of extraction site (ridge) [Mean (Standard Deviation); unit: mm] | 13.7 (1.2) | 13 (1.96) | 13.36 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Width of Extraction Site (Ridge)
Description: the distance from the buccal plate to the palatal plate
Time Frame: 8 months
Population: A total of six participants (four females and two males) completed this pilot study. Their mean age was 37 ± 21 years (range, 22-68).
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Teeth
Arm/Group | Mini-screw Placement | No Treatment
Number analyzed (Participants) | 3 | 3
Number analyzed (Teeth) | 6 | 6
mm | 0.7 (0.2) | 1.3 (0.7)
Statistical Analysis 1: Comparison: Mini-screw Placement vs No Treatment; Test type: Superiority; p < 0.05, Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- No Treatment: No treatment after tooth extraction
Arm/Group | Mini-screw Placement | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mini-screw Placement (N=3) | No Treatment (N=3)
Inflammation at site (Infections and infestations) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03205800/Prot_SAP_001.pdf